CLINICAL TRIAL: NCT00199394
Title: A 16-week, Double-Blind, Placebo-Controlled, Randomised, Parallel-Group, Multicentre, International Study to Evaluate the Efficacy and Safety of 40 mg/Day KW-6002 (Istradefylline) and That of Entacapone Versus Placebo as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa Therapy.
Brief Title: A Study of Istradefylline (KW-6002) for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin UK, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-EU-007
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: KW-6002 (istradefylline); Entacapone; Placebo; Parkinson's Disease; Motor Response Complications; Levodopa Therapy
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
The purpose of this study is to evaluate the efficacy of 40 mg a day of istradefylline (KW-6002) for reducing the percentage of awake time spent in the OFF state in patients with advanced Parkinson's disease treated with levodopa.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive motor disease characterized by bradykinesia or akinesia, rigidity, and resting tremor. Levodopa is still the most widely used treatment for PD, but as the disease progresses the drug tends to become less helpful. This is because of the development of motor response complications such as end-of-dose deterioration or wearing-off, peak dose dyskinesias, and ON-OFF phenomenon.

Comparison(s): The safety of 40 mg/d istradefylline and the efficacy for reducing the percentage of OFF time in patients with advanced PD treated with levodopa will be compared to placebo. The safety and efficacy of Entacapone will also be compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients selected for this study will be at least 30 years of age and will have been diagnosed with advanced Parkinson's disease as determined by UK Parkinson's Disease Society (UKPDS) criteria and the Modified Hoehn and Yahr Scale. The patients will have been receiving levodopa treatment for at least one year, may be taking other antiparkinsonian drugs, will have an average of at least three hours OFF time as recorded in two 24-hour ON/OFF diaries, and if female, must be non-pregnant and non-nursing.

Exclusion Criteria:

Patients may not be enrolled if they are taking certain medications excluded by the protocol, have been treated with any investigational drug within 30 days prior to randomisation (or five half-lives if longer), have ever received istradefylline or been treated with a COMT inhibitor, are psychotic, have clinically significant illness or laboratory values at screening, have insufficient mental capacity to comply with protocol requirements or certain psychiatric or neurological conditions.

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405
Dates: Start 2004-11; Primary Completion 2005-10 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
OFF time assessed by patient diaries at endpoint.

SECONDARY OUTCOMES:
Efficacy: OFF time
ON time
UPDRS (parts I-IVa)
PDQ-39, PCG-I, CGI-S and SF-36 scores at endpoint.
Safety: clinical laboratory tests
12-lead ECG
vital signs
physical (including neurological) examination and adverse events throughout.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyowa Hakko UK Ltd., Slough, Berkshire, United Kingdom